CLINICAL TRIAL: NCT00843102
Title: Investigation of Coronary and Pulmonary Circulatory Parameters in Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, András Komócsi, senior lecturer, University of Pecs
Other Study IDs: 330/PI/2007
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Systemic Sclerosis
Keywords: atherosclerosis; pulmonary hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Atherosclerosis; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim: Determination of frequency and nature of coronary involvement (including epicardial and microvascular) among scleroderma patients referred for right heart catheterization.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc)is a multiorgan autoimmune disease characterized by fibrosis of the skin and internal organs. Cardio-pulmonary manifestation in systemic sclerosis (SSc) patients has significant impact on the prognosis. Several elements of the heart and lung involvement encountered frequently in combination. Clinically apparent SSc cardiac involvement is recognized as poor prognostic factor, and in our experience it is the most frequent cause of death among SSc patients. Moreover arrhythmias, diastolic and less frequently systolic dysfunction considerably interfere with the quality of life of these patients. Cardiac involvement includes primary cardiac disorders like fibrosis of the contractile elements, ischemia due to the involved microcirculation and/or to the epicardial coronaries and some secondary ones like consequences of systemic or pulmonary hypertension.

Autopsy identifies fibrosis of the myocardium in up to 80 percent of cases. Its distribution is unrelated to epicardial coronary stenosis, and inflammatory processes are thought to play substantial role in its evolution. Microvascular disease (MVD) that causes reduction of the vasodilatory capacity independently from epicardial coronary disease (CAD), is known for several decades. Short term benefits from vasodilatory treatment has been also reported in some latest studies.

Symptoms of the elements of cardio-pulmonary involvement overlap and coronary abnormalities alike MVD were also found in asymptomatic patients. Recently prevalence of CAD is reported to be similar to gender, age and symptom matched controls. Atypical clinical presentations were predominant and nevertheless these findings indicate that SSc patients are not free from CAD.

Clarification the causes of reduced exercise capacity, chest pain and faint in SSc is a challenging task and requires multidisciplinary approach. Driven by its high mortality and due to the recent emergence of effective therapy SSc patients are regularly screened for pulmonary hypertension (PAH). Clinical presentation of scleroderma related PAH is unspecific. Fatigue, chest pain and dyspnea may be related to other organs, such as the lung, musculoskeletal system or the esophagus. The definitive diagnosis of PAH still depends on the results of right heart catheterization (RHC). As the non-invasive diagnostics are influenced and to some extent restricted by multiple clinical manifestations, RHC is performed liberally in symptomatic patients. Still a considerable proportion of patients who underwent RHC have normal pulmonary pressure and the cause of symptoms may remain obscure as cardiac involvement may not be correctly diagnosed or entirely overlooked.

We intend to characterize coronary artery disease in symptomatic SSc patients by means of a prospective cross-sectional study consisting of organized screening of SSc patients and systematic left heart catheterization (coronary angiography, and coronary flow reserve estimation) in all patients referred to RHC. Prognostic impact of the different manifestations are determined during five-year follow-up of the study.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatologist established systemic sclerosis
* informed consent

Exclusion Criteria:

* left ventricular ejection fraction <30%
* severly (<60% of predicted) deteriorated pulmonary function

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Systemic sclerosis
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of angiography proven coronary disease | 1 year
Occurence of pulmonary arterial hypertension | 1 year

SECONDARY OUTCOMES:
Overall mortality | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pécs, Hungary, Pécs, Hungary

REFERENCES:
- [Result] Komocsi A, Pinter T, Faludi R, Magyari B, Bozo J, Kumanovics G, Minier T, Radics J, Czirjak L. Overlap of coronary disease and pulmonary arterial hypertension in systemic sclerosis. Ann Rheum Dis. 2010 Jan;69(1):202-5. doi: 10.1136/ard.2008.096255. PMID 19158116
- [Derived] Kolto G, Faludi R, Aradi D, Bartos B, Kumanovics G, Minier T, Czirjak L, Komocsi A. Impact of cardiac involvement on the risk of mortality among patients with systemic sclerosis: a 5-year follow-up of a single-center cohort. Clin Rheumatol. 2014 Feb;33(2):197-205. doi: 10.1007/s10067-013-2358-4. Epub 2013 Aug 14. PMID 23942767